CLINICAL TRIAL: NCT04521816
Title: PIM 2.0: Patient Aligned Care Team (PACT) Intensive Management (PIM) Project
Acronym: PIM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veteran Affairs Office of Patient Care Services (U.S. Federal Agency)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PIM #2
Record Dates: First submitted 2020-07-08; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Primary Health Care; Health Care Costs
Keywords: High-Risk Patients, Complex patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention--PACT Intensive Management (Experimental): The intervention is the PACT Intensive Management Program (PIM) provides a standardized menu of services, ranging from chart review assessment or in-home assessment, to a time limited intensive care management intervention. The following PIM features are standardized across the PIM demonstration sites:
  A) Chart review assessment template in the EMR; B) Comprehensive assessment template of unmet needs and modifiable risk factors in EMR; C) Transitions in care process (eligibility criteria, clinical protocols); D) Diagnostic home visits process (eligibility criteria, clinical protocols); E) Core risk stratification/Triage process; F) Discharge criteria and note template in EMR; G) Standardized interdisciplinary team (IDT) meeting note procedure and template in EMR.
  Interventions: Behavioral: PACT Intensive Management
- Usual care (No Intervention): High-Risk patients receiving care in PACT.

INTERVENTIONS:
Behavioral: PACT Intensive Management — Purpose: Implement a Patient Aligned Care Team (PACT) model that identifies and proactively manages Veterans at the highest risk for hospital admission and death while they are still in the ambulatory care setting.
  Goal:
  * Reduce emergency department and urgent care utilization, hospitalization, and mortality in complex, high risk patients
  * Improve Veteran and staff satisfaction
  Objectives:
  * Maintain the patient in the home setting as much as possible
  * Secure appropriate home environment to facilitate health and well-being
  * Utilize comprehensive team-based care
  * Engage appropriate VHA programs to provide interdisciplinary, coordinated, and timely management of complex medical issues
  Other Names: PIM
  Arms: Intervention--PACT Intensive Management

SUMMARY:
Purpose: Implement a Patient Aligned Care Team (PACT) model that identifies and proactively manages Veterans at the highest risk for hospital admission and death while the patient is still in the ambulatory care setting.

Goal:

* Reduce emergency department and urgent care utilization, hospitalization, and mortality in complex, high risk patients
* Improve Veteran and staff satisfaction

Objectives:

* Maintain the patient in the home setting as much as possible
* Secure appropriate home environment to facilitate health and well-being
* Utilize comprehensive team-based care
* Engage appropriate Veteran Health Administration (VHA) programs to provide interdisciplinary, coordinated, and timely management of complex medical issues

ELIGIBILITY:
Inclusion Criteria:

* Refered for intensive management

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
VA health care cost | 2 years (two 1-year points)
  Total costs of VA care, including inpatient, outpatient, pharmacy and fee-basis services.

SECONDARY OUTCOMES:
Healthcare Utilization | 2 years (two 1-year points)
  VA central repository administrative data will be analyzed to calculate utilization of hospital, emergency and outpatient primary and specialty care. This information will be electronically abstracted through the VA central repository administrative data center
Total Medicare Cost | 2 years (two 1-year points)
  Data will be extracted from VHA's Corporate Data Warehouse to capture patient Medicare cost. Medicare claims data to measure total patient inpatient and outpatient cost for services reimbursed by Medicare. Inpatient cost will be measured as cost for total acute hospitalizations, and subcategories: medical, surgical, psychiatric, rehabilitation, hospice and ambulatory care-sensitive conditions. Outpatient cost will be measured as the cost for combined visits in VHA and elsewhere reimbursed by Medicare in 9 categories: primary care, specialty care, mental health, surgical, home health, nursing home, diagnostic, rehabilitation and ED.
Total Medicare Utilization | 2 years (two 1-year points)
  Data will be extracted from VHA's Corporate Data Warehouse to capture patient utilization. Medicare claims data to measure total patient inpatient and outpatient utilization for services reimbursed by Medicare. Inpatient utilization will be measured as counts of total acute hospitalizations, and subcategories: medical, surgical, psychiatric, rehabilitation, hospice and ambulatory care-sensitive conditions. Outpatient utilization will be measured as the number of combined visits in VHA and elsewhere reimbursed by Medicare in 9 categories: primary care, specialty care, mental health, surgical, home health, nursing home, diagnostic, rehabilitation and ED.

OTHER OUTCOMES:
Functional status- General | 2 years (two 1-year points)
  Patient report of their physical, social, and mental functional status is routinely collected as part of their medical visit as health factor data. The data will be abstracted through the VA central repository administrative data. The variables used to measure functional status are the following:
  •In general, please rate how well you carry out your usual social activities and roles. (This includes activities at home, at work and in your community, and responsibilities as a parent, child, spouse, employee, friend, etc.) (Excellent, Very good, Good, Fair, Poor)
Functional Status- Social | 2 years (two 1-year points)
  Patient report of their physical, social, and mental functional status is routinely collected as part of their medical visit as health factor data. The data will be abstracted through the VA central repository administrative data. The variables used to measure functional status are the following:
  •In general, how would you rate your satisfaction with your social activities and relationships? (Excellent, Very good, Good, Fair, Poor)
Functional status- ADLS | 2 years (two 1-year points)
  Patient report of their physical, social, and mental functional status is routinely collected as part of their medical visit as health factor data. The data will be abstracted through the VA central repository administrative data. The variables used to measure functional status are the following:
  •Administer Katz Index of Independence in Activities of Daily Living (Independence=1 point; dependence = 0 points for each of the six item pairs)
Functional status- IDLS | 2 years (two 1-year points)
  Patient report of their physical, social, and mental functional status is routinely collected as part of their medical visit as health factor data. The data will be abstracted through the VA central repository administrative data. The variables used to measure functional status are the following:
  •Administer the Lawton Instrumental Activities of Daily Living (IADL) Scale (score 0-8)
Patient Quality of Life Status | 2 years (two 1-year points)
  Patient assessment of their quality of life collected as part of their medical care as a health factor. This information will be electronically abstracted through the VA central repository administrative data center. The variables used to assess a patient's quality of life are the following:
  * Patient's self-rating of quality of life in general: Excellent, Very Good, Good, Fair, Poor
  * Patient's self-rating of mental health, including mood and ability to think: Excellent, Very Good, Good, Fair, Poor
Patient Symptom Burden | 2 years (two 1-year points)
  Patient assessment of symptom burden is routinely collected as part of their care and documented in their medical record and will be electronically abstracted through the VA central repository administrative data center. Mental Health and physical burdens are abstracted from the medical record utilizing ICD-9 and ICD-10 code. It will be assessed as yes/no if present.
Anxiety | 2 years (two 1-year points)
  Generalized Anxiety Disorder 2-item (GAD-2): (Not at all; several days; More than half the days, nearly every day). The higher the score the higher the anxiety.
Substance Abuse | 2 years (two 1-year points)
  The 3-item AUDIT-C scored on a scale of 0-12; Drugs: How many times in the past year, have you used an illegal drug or used a prescription medication for nonmedical reasons? (Yes/No, Number of times). The greater the score the worse the substance abuse status.
Cognitive Status | 2 years (two 1-year points)
  The Blessed-Short and/or the Mini-Cog where the lower the score the more impairment.
Pain level | 2 years (two 1-year points)
  Pain in past 24 hours on scale of 0 = no pain, to 10 = worst pain imaginable.
Shortness of Breath | 2 years (two 1-year points)
  Shortness of breath in past 24 hours on a scale of 0, no shortness of breath, to 10, worst imaginable.
Problems with constipation | 2 years (two 1-year points)
  Constipation in past 24 hours on a scale from 0, no constipation, to 10, worst imaginable.
Sleep Problems | 2 years (two 1-year points)
  Sleep problems in past 24 hours on a scale from 0, no sleep problems, to 10, worst imaginable.
Level of Fatigue | 2 years (two 1-year points)
  Fatigue in past 24 hours on a scale from 0, no fatigue, to 10, worst imaginable.
Risk of Falls | 2 years (two 1-year points)
  Falls (Patient reports no falls in past 12 months;Patient reports no problems with walking or balance; Patient reports problems with walking or balance; Patients reports falls in past 12 months
Patient Satisfaction-Trust | 2 years (two 1-year points)
  I have a VA healthcare provider who I can trust. 1: Very dissatisfied 2: Dissatisfied 3: Somewhat dissatisfied 4: Somewhat satisfied 5: Satisfied 6: Very satisfied
Patient Satisfaction- Care Coordination | 2 years (two 1-year points)
  I have a VA healthcare provider who helps coordinate my care from different doctors and services. 1: Very dissatisfied 2: Dissatisfied 3: Somewhat dissatisfied 4: Somewhat satisfied 5: Satisfied 6: Very satisfied
Patient Satisfaction- Access | 2 years (two 1-year points)
  I got the service I needed. 1: Very dissatisfied 2: Dissatisfied 3: Somewhat dissatisfied 4: Somewhat satisfied 5: Satisfied 6: Very satisfied
Patient Satisfaction- Goals | 2 years (two 1-year points)
  In the last 6 months, did someone at the VA talk with you about specific goals for your health. 1: Very dissatisfied 2: Dissatisfied 3: Somewhat dissatisfied 4: Somewhat satisfied 5: Satisfied 6: Very satisfied
Patient Satisfaction- Help with Barriers | 2 years (two 1-year points)
  In the last 6 months, did someone at the VA ask you if there are things that make it hard for you to take care of your health. 1: Very dissatisfied 2: Dissatisfied 3: Somewhat dissatisfied 4: Somewhat satisfied 5: Satisfied 6: Very satisfied
Patient Satisfaction- overall facility | 2 years (two 1-year points)
  Overall, how satisfied are you with the health care you have received at your VA facility?
  1. Very dissatisfied
  2. Dissatisfied
  3. Somewhat dissatisfied
  4. Somewhat satisfied
  5. Satisfied
  6. Very satisfied
Patient Satisfaction- overall provider | 2 years (two 1-year points)
  is the best provider possible, what number would you use to rate this provider?
  1. Very dissatisfied
  2. Dissatisfied
  3. Somewhat dissatisfied
  4. Somewhat satisfied
  5. Satisfied
  6. Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Chang, MD, Principal Investigator — VAGLAHS- WLA
Locations (1):
- VAGLAHS, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang ET, Huynh A, Yoo C, Yoon J, Zulman DM, Ong MK, Klein M, Eng J, Roy S, Stockdale SE, Jimenez EE, Denietolis A, Needleman J, Asch SM; PACT Intensive Management (PIM) Demonstration Sites, PIM National Evaluation Center, and PIM Executive Committee. Impact of Referring High-Risk Patients to Intensive Outpatient Primary Care Services: A Propensity Score-Matched Analysis. J Gen Intern Med. 2025 Feb;40(3):637-646. doi: 10.1007/s11606-024-08923-3. Epub 2024 Jul 29. PMID 39075268

DOCUMENTS (1):
  • Study Protocol (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT04521816/Prot_000.pdf